CLINICAL TRIAL: NCT00901836
Title: A Pilot Study Investigating Preoperative Proton Radiotherapy for Retroperitoneal Sarcoma
Brief Title: Preoperative Proton Radiotherapy for Retroperitoneal Sarcoma
Acronym: SA03
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to feasability
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0805-SA03
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Retroperitoneal Sarcoma
Keywords: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Proton Therapy (Experimental): 28 daily fractions of 1.8 cobalt gray equivalent(CGE)/fx for total of 50.4 CGE over 5.5 weeks.
  Interventions: Radiation: Preoperative proton therapy
- Surgery (Active Comparator): Standard of care surgery will be performed 4-6 weeks after the completion of radiation.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Radiation: Preoperative proton therapy — 28 daily fractions of 1.8 cobalt gray equivalent(CGE)/fx for total of 50.4 CGE over 5.5 weeks.
  Arms: Preoperative Proton Therapy
Procedure: Surgery — Standard of care surgery will be performed 4-6 weeks after completion of radiation.
  Arms: Surgery

SUMMARY:
The goal of this study is to evaluate radiation treatment intended to increase the chance of curing your sarcoma and decrease the side effects of proton therapy.

This study will also look at the tumor tissue that was removed during your initial biopsy and your final surgery for information that may help to treat retroperitoneal sarcoma in the future.

DETAILED DESCRIPTION:
Data collection will be obtained from the patient's medical records including initial evaluation, pathology report, dosimetry information, radiotherapy completion records and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed intermediate or high grade retroperitoneal sarcomas of any histologic subtype.
* Primary or recurrent disease isolated to a single intra-abdominal or retroperitoneal region is allowed.
* Tumor must be considered potentially completely resectable as defined by cross sectional imaging (no 360o encasement of the superior mesenteric artery, aorta, inferior vena cava, iliac arteries or iliac veins and no extension of tumor into the vertebral column).
* At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have ≤ grade 1 acute toxicities of any prior treatment with anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤ grade 1 are eligible.
* Age ≥18 years at time of consent.
* Life expectancy of greater than 3 months. Physician documented.
* Women of child-producing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and the subsequent 6 months. Patients must have a negative serum pregnancy test within 2 weeks prior to beginning treatment on this trial. Sexually active men must also use appropriate contraception method and should not father a child while receiving therapy during this study.
* Ability to understand and the willingness to sign a written Institutional Review Board(IRB) stamped study specific informed consent document before undergoing research related procedures or study treatment.
* Biopsy is required with pathologic confirmation of intermediate or high grade sarcoma with pathology review at the University of Florida.
* Agree to allow their tissue to be used for current study.

Exclusion Criteria:

* Receiving any investigational agents.
* Evidence of metastatic disease.
* Uncontrolled intercurrent illness and/or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded from this study because the radiotherapy may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated.
* All herbal and/or alternative medications should be discontinued while on study, including, but not limited to: Hydrastis canadensis (goldenseal), Uncaria tomentosa (cat's claw) or Echinacea angustifolia.
* Requirement for treatment with immunosuppressive agents or chronic steroids.
* Previous intra-abdominal or retroperitoneal radiotherapy.
* Treatment with cytotoxic agents and/or treatment with biologic agents within the 4 weeks prior to beginning treatment on this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To assess treatment feasibility of preoperative proton therapy for resectable intermediate or high grade retroperitoneal sarcoma. | 4-6 weeks post treatment

SECONDARY OUTCOMES:
To evaluate the acute and late toxicity of preoperative proton therapy for resectable intermediate or high grade retroperitoneal sarcoma | Weekly during treatment, then every 3 months for 1 year, then every 6 months for 4 years.
To determine the incidence of margin negative resection in patients compared to historic controls treated with photon therapy. | 4-6 weeks post treatment
To determine the percent tumor necrosis and percent apoptosis compared to historic controls treated with photon therapy. | 4-6 weeks post treatment
To assess the predictive value of CT and MRI in evaluating pathologic tumor response and margin negative resection following proton radiotherapy. | 4-6 weeks post treatment
To compare the dose distribution to tumor and surrounding normal structures using dose volume histograms (DVHs) generated from the proton plan used to treat the patient and a theoretical photon plan generated for comparison purposes. | 4-6 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Indelicato, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaques DP, Coit DG, Hajdu SI, Brennan MF. Management of primary and recurrent soft-tissue sarcoma of the retroperitoneum. Ann Surg. 1990 Jul;212(1):51-9. doi: 10.1097/00000658-199007000-00008. PMID 2363604
- [Background] Ferrario T, Karakousis CP. Retroperitoneal sarcomas: grade and survival. Arch Surg. 2003 Mar;138(3):248-51. doi: 10.1001/archsurg.138.3.248. PMID 12611567
- [Background] Heslin MJ, Lewis JJ, Nadler E, Newman E, Woodruff JM, Casper ES, Leung D, Brennan MF. Prognostic factors associated with long-term survival for retroperitoneal sarcoma: implications for management. J Clin Oncol. 1997 Aug;15(8):2832-9. doi: 10.1200/JCO.1997.15.8.2832. PMID 9256126
- [Background] Lewis JJ, Leung D, Woodruff JM, Brennan MF. Retroperitoneal soft-tissue sarcoma: analysis of 500 patients treated and followed at a single institution. Ann Surg. 1998 Sep;228(3):355-65. doi: 10.1097/00000658-199809000-00008. PMID 9742918
- [Background] Kilkenny JW 3rd, Bland KI, Copeland EM 3rd. Retroperitoneal sarcoma: the University of Florida experience. J Am Coll Surg. 1996 Apr;182(4):329-39. PMID 8605556
- [Background] Lewis JJ, Brennan MF. The management of retroperitoneal soft tissue sarcoma. Adv Surg. 1999;33:329-44. No abstract available. PMID 10572575
- [Background] Harrison LB, Gutierrez E, Fischer JJ. Retroperitoneal sarcomas: the Yale experience and a review of the literature. J Surg Oncol. 1986 Jul;32(3):159-64. doi: 10.1002/jso.2930320309. PMID 3736052
- [Background] van Doorn RC, Gallee MP, Hart AA, Gortzak E, Rutgers EJ, van Coevorden F, Keus RB, Zoetmulder FA. Resectable retroperitoneal soft tissue sarcomas. The effect of extent of resection and postoperative radiation therapy on local tumor control. Cancer. 1994 Feb 1;73(3):637-42. doi: 10.1002/1097-0142(19940201)73:33.0.co;2-y. PMID 8299085
- [Background] Tepper JE, Gunderson LL, Orlow E, Cohen AM, Hedberg SE, Shipley WU, Blitzer PH, Rich T. Complications of intraoperative radiation therapy. Int J Radiat Oncol Biol Phys. 1984 Oct;10(10):1831-9. doi: 10.1016/0360-3016(84)90258-x. PMID 6436198
- [Background] Koshy M, Landry JC, Lawson JD, Staley CA, Esiashvili N, Howell R, Ghavidel S, Davis LW. Intensity modulated radiation therapy for retroperitoneal sarcoma: a case for dose escalation and organ at risk toxicity reduction. Sarcoma. 2003;7(3-4):137-48. doi: 10.1080/13577140310001644751. PMID 18521378
- [Background] Weber DC, Rutz HP, Bolsi A, Pedroni E, Coray A, Jermann M, Lomax AJ, Hug EB, Goitein G. Spot scanning proton therapy in the curative treatment of adult patients with sarcoma: the Paul Scherrer institute experience. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):865-71. doi: 10.1016/j.ijrobp.2007.04.034. Epub 2007 Jul 2. PMID 17606333
- [Background] Zlotecki RA, Katz TS, Morris CG, Lind DS, Hochwald SN. Adjuvant radiation therapy for resectable retroperitoneal soft tissue sarcoma: the University of Florida experience. Am J Clin Oncol. 2005 Jun;28(3):310-6. doi: 10.1097/01.coc.0000158441.96455.31. PMID 15923806
- [Background] Tuma RS. Sometimes size doesn't matter: reevaluating RECIST and tumor response rate endpoints. J Natl Cancer Inst. 2006 Sep 20;98(18):1272-4. doi: 10.1093/jnci/djj403. No abstract available. PMID 16985244
- [Background] Pollack A, Zagars GK, Goswitz MS, Pollock RA, Feig BW, Pisters PW. Preoperative vs. postoperative radiotherapy in the treatment of soft tissue sarcomas: a matter of presentation. Int J Radiat Oncol Biol Phys. 1998 Oct 1;42(3):563-72. doi: 10.1016/s0360-3016(98)00277-6. PMID 9806516
- [Background] Suit HD, Mankin HJ, Wood WC, Proppe KH. Preoperative, intraoperative, and postoperative radiation in the treatment of primary soft tissue sarcoma. Cancer. 1985 Jun 1;55(11):2659-67. doi: 10.1002/1097-0142(19850601)55:113.0.co;2-q. PMID 3995476
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Davis AM, O'Sullivan B, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Hammond A, Benk V, Kandel R, Goddard K, Freeman C, Sadura A, Zee B, Day A, Tu D, Pater J; Canadian Sarcoma Group; NCI Canada Clinical Trial Group Randomized Trial. Late radiation morbidity following randomization to preoperative versus postoperative radiotherapy in extremity soft tissue sarcoma. Radiother Oncol. 2005 Apr;75(1):48-53. doi: 10.1016/j.radonc.2004.12.020. PMID 15948265
- [Background] Borden EC, Baker LH, Bell RS, Bramwell V, Demetri GD, Eisenberg BL, Fletcher CD, Fletcher JA, Ladanyi M, Meltzer P, O'Sullivan B, Parkinson DR, Pisters PW, Saxman S, Singer S, Sundaram M, van Oosterom AT, Verweij J, Waalen J, Weiss SW, Brennan MF. Soft tissue sarcomas of adults: state of the translational science. Clin Cancer Res. 2003 Jun;9(6):1941-56. PMID 12796356
- [Background] Baglan KL, Frazier RC, Yan D, Huang RR, Martinez AA, Robertson JM. The dose-volume relationship of acute small bowel toxicity from concurrent 5-FU-based chemotherapy and radiation therapy for rectal cancer. Int J Radiat Oncol Biol Phys. 2002 Jan 1;52(1):176-83. doi: 10.1016/s0360-3016(01)01820-x. PMID 11777636
- [Background] Robertson JM, Lockman D, Yan D, Wallace M. The dose-volume relationship of small bowel irradiation and acute grade 3 diarrhea during chemoradiotherapy for rectal cancer. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):413-8. doi: 10.1016/j.ijrobp.2007.06.066. Epub 2007 Sep 27. PMID 17904305
- [Background] Letschert JG. The prevention of radiation-induced small bowel complications. Eur J Cancer. 1995 Jul-Aug;31A(7-8):1361-5. doi: 10.1016/0959-8049(95)00179-m. PMID 7577052
- [Background] Sindelar WF, Kinsella TJ, Chen PW, DeLaney TF, Tepper JE, Rosenberg SA, Glatstein E. Intraoperative radiotherapy in retroperitoneal sarcomas. Final results of a prospective, randomized, clinical trial. Arch Surg. 1993 Apr;128(4):402-10. doi: 10.1001/archsurg.1993.01420160040005. PMID 8457152